CLINICAL TRIAL: NCT04300010
Title: Efficacy of Blue Light Therapy in Reducing Cutibacterium Acnes Bioburden at the Deltopectoral Interval
Brief Title: Blue Light Therapy of C. Acnes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0018; A536110 (Other: UW Madison); SMPH/ORTHO&REHAB/ORTHO (Other: UW Madison); Protocol Version 9/14/2020 (Other: UW Madison)
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Phototherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Blue Light Therapy (Active Comparator): FDA cleared blue light product, Omniluxblue (Globalmed Technologies, Glen Elen, CA), which emits a 415 nm blue light irradiance of 40mW/cm2. Following the application of blue light protective eyewear, the blue light therapy device will be centered over the deltopectoral interval according to device standardized use instructions and a 23-minute treatment will be administered to dry skin. As was done in the topical BPO group, following treatment, a skin swab culture of the treatment shoulder will be taken, then both the treatment shoulder and control shoulder will be sterilely prepped with 2% chlorhexidine gluconate solution with 70% isopropyl alcohol and allowed to dry for 3 minutes. Following chlorhexidine preparation, a single set of cultures will be obtained from each shoulder. Participants and research personnel conducting the blue light treatments will be wearing medical grade blue light protective glasses for safety.
  Interventions: Device: Blue Light Therapy
- 5% Topical Benzoyl Peroxide Gel (Active Comparator): A pea-sized amount, ~0.5 grams, will be applied to a 10cm strip over the deltopectoral interval beginning the morning 48 hours prior to schedule research visit to obtain cultures. The benzoyl peroxide will be applied on dry skin after a shower. The gel will be applied once in the morning and once in the evening for two consecutive days as well as the morning of the scheduled research visit. Following treatment, a skin swab culture of the treatment shoulder will be taken, both the treatment shoulder and control shoulder will be sterilely prepped with 2% chlorhexidine gluconate solution with 70% isopropyl alcohol and allowed to dry for 3 minutes. Following chlorhexidine preparation, a single set of cultures will be obtained from each shoulder.
  Interventions: Drug: 5% Topical Benzoyl Peroxide Gel
- Light and Gel (Active Comparator): Prior to treatment, a skin swab culture will be taken, 5% topical benzoyl peroxide treatment will be performed on dry skin immediately after a shower as described in the above paragraph. Again, five total treatments will be performed prior to research visit. On the day of the research visit, the blue light therapy protocol described above will be performed exactly the same followed by culture obtainment.
  Interventions: Drug: 5% Topical Benzoyl Peroxide Gel; Device: Blue Light Therapy

INTERVENTIONS:
Drug: 5% Topical Benzoyl Peroxide Gel — Gel treatment used to treat acne
  Arms: 5% Topical Benzoyl Peroxide Gel; Light and Gel
Device: Blue Light Therapy — Blue light therapy treatment for acne
  Arms: Blue Light Therapy; Light and Gel

SUMMARY:
This proposal aims to investigate a novel light-based treatment to reduce morbidity in shoulder surgical patients. This has potential to improve outcomes and reduce health care utilization associated with infectious complications of shoulder arthroplasty. Participants will be healthy male volunteers at least 18 years of age. They will be on study for approximately 2 days.

DETAILED DESCRIPTION:
Participants will have two study visits (consent plus treatment and swabs for culture). These visits will be conducted at the main UW Hospital, UW Health at the American Center, or UW Health at 1 S. Park. All visits will be conducted in reserved conference rooms at each location.

Once a subject is determined to be eligible and has consented to the study, they will be randomized into one of three treatment groups. Study team has blank envelopes that contain one of the three treatment groups enclosed. After a subject consents to the study, the study team will randomly draw an envelope to assign a treatment arm.

Arm 1. One group will receive 5% topical benzoyl peroxide gel plus 2% chlorhexidine gluconate with 70% isopropyl alcohol

Arm 2. One group will receive blue light therapy plus 2% chlorhexidine gluconate with 70% isopropyl alcohol

Arm 3. One group will receive both of the above treatments

All participants will have their contralateral shoulder serve as the control (2% chlorhexidine gluconate with 70% isopropyl alcohol only). All treatment will be provided by the study team. Participants will also be asked to complete a research intake form.

If C. acnes does grow for a tissue culture, Investigators plan to bank a colony of the bacterium for potential use in a future study. There will be no added risk to research subjects as no additional cultures will be taken and samples will be completely anonymized. The banked samples will simply be a colony of growth from the culture media for storage for possible future use. Samples will be banked for 5 years from the date of study completion after which time the samples will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* 18 years or older

Exclusion Criteria:

* Allergy to benzoyl peroxide or chlorhexidine
* <18 years of age
* Previous history of shoulder infections
* Antibiotics taken within one month of research visit
* Immunocompromised state
* Active cancer
* Diabetic
* Skin lesions or abrasions over the deltopectoral interval
* Topical corticosteroid treatment to either shoulder or or systemic corticosteroid treatment within 2 weeks of research visit
* Topical benzoyl peroxide treatment to either shoulder within 2 weeks of research visit
* Blue light therapy treatment to either shoulder within 2 weeks of research visit
* Prior incision over the deltopectoral interval of either shoulder
* Contraindication to blue light treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males have a higher incidence of C. Acnes. Inclusion criteria includes males 18 years of age and older, as this is the gender and age group most likely to have C. Acnes.
Enrollment: 60 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian F Grogan, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cotter EJ, Cotter LM, Franczek EB, Godfrey JJ, Hetzel SJ, Safdar N, Dai T, Arkin L, Grogan BF. Efficacy of combinational therapy using blue light and benzoyl peroxide in reducing Cutibacterium acnes bioburden at the deltopectoral interval: a randomized controlled trial. J Shoulder Elbow Surg. 2021 Dec;30(12):2671-2681. doi: 10.1016/j.jse.2021.08.008. Epub 2021 Aug 31. PMID 34478863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited through fliers around the study institution's facilities, through Clinicaltrials.gov, and informational emails to clinical staff listservs at the study University of Wisconsin - Madison. Participants were enrolled from 10/5/20 through 1/22/21.
Units Other Than Participants: shoulders
Groups:
- Blue Light Therapy: The blue light therapy device will be centered over the deltopectoral interval according to device standardized use instructions and a 23-minute treatment will be administered to dry skin. Following treatment, a skin swab culture of the treatment shoulder will be taken, then both the treatment shoulder and control shoulder will be sterilely prepped with 2% chlorhexidine gluconate solution with 70% isopropyl alcohol and allowed to dry for 3 minutes. Following chlorhexidine preparation, a single set of cultures will be obtained from each shoulder.
- Control Shoulder: All participants will have their contralateral shoulder serve as the control (2% chlorhexidine gluconate with 70% isopropyl alcohol only)
Period: Overall Study
Arm/Group | Blue Light Therapy | 5% Topical Benzoyl Peroxide Gel | Light and Gel | Control Shoulder
Started | 20; 20 shoulders | 20; 20 shoulders | 20; 20 shoulders | 60; 60 shoulders
Completed | 20; 20 shoulders | 20; 20 shoulders | 20; 20 shoulders | 60; 60 shoulders
Not Completed | 0; 0 shoulders | 0; 0 shoulders | 0; 0 shoulders | 0; 0 shoulders

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blue Light Therapy | 5% Topical Benzoyl Peroxide Gel | Light and Gel | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.70 (2.99) | 26.80 (3.62) | 25.90 (2.97) | 26.47 (2.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 20 | 20 | 20 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 19 | 19 | 18 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 3 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 1 | 0 | 2
  White | 13 | 14 | 15 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.60 (3.49) | 24.56 (2.30) | 24.63 (3.92) | 24.60 (3.67)
Occupation [Count of Participants; unit: Participants]
  Student | 15 | 13 | 16 | 44
  Resident | 5 | 7 | 3 | 15
  Other Healthcare Professional | 0 | 0 | 1 | 1
Asthma [Count of Participants; unit: Participants] | 2 | 3 | 0 | 5
Autoimmune Condition [Count of Participants; unit: Participants] | 0 | 0 | 2 | 2
Infection Requiring Intravenous Antibiotics [Count of Participants; unit: Participants] | 1 | 0 | 1 | 2
Consume Alcohol [Count of Participants; unit: Participants] | 18 | 16 | 19 | 53
Number of Alcohol Drinks per Week [Mean (Standard Deviation); unit: drinks per week] — One drink is 1 12oz beer, 5 ounces of wine, or 1.5 ounces of distilled spirits per the NIH definition.
  drinks per week | 2.05 (1.78) | 2.15 (1.91) | 2.58 (2.01) | 2.26 (1.89)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With C. Acnes Bacterium Culture After Treatment
Description: Swab will be taken from skin and cultured for approximately 7 days to determine bacteria growth. This result is for the null condition following treatment with either blue light, blue light plus benzoyl peroxide or just benzoyl peroxide but before additional preparation with chlorhexidine.
Time Frame: up to 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Blue Light Therapy | 5% Topical Benzoyl Peroxide Gel | Light and Gel
Number analyzed (Participants) | 20 | 20 | 20
Participants | 20 | 20 | 16

2. Primary Outcome: Median Colony Forming Units (CFU) After Treatment
Description: Quantitative culture analysis between treatment groups after treatment to the shoulder but before chlorhexidine preparation (null condition).
Time Frame: up to 2 days
Measure: Median (Inter-Quartile Range); unit: CFU/mL
Arm/Group | Blue Light Therapy | 5% Topical Benzoyl Peroxide Gel | Light and Gel
Number analyzed (Participants) | 20 | 20 | 20
CFU/mL | 304000 [77800 to 915000] | 28500 [10300 to 89000] | 12100 [300 to 143000]

3. Primary Outcome: Percentage of Participants in Each Group With Positive C. Acnes Cultures
Description: Comparison of positive Cutibacterium acnes cultures as a binary (yes/no) outcome between treatment arm and control arm following chlorhexidine (CHX) prep. Reported is the percentage of people in each group that had Cutibacterium acnes growth.
Time Frame: up to 2 days
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Blue Light Therapy | 5% Topical Benzoyl Peroxide Gel | Light and Gel
Number analyzed (Participants) | 20 | 20 | 20
percent
  Treatment plus CHX Arm | 90.0 [67.6 to 97.5] | 15.0 [4.9 to 37.6] | 40.0 [21.4 to 62.0]
  Control Arm after CHX | 80.0 [57.2 to 92.3] | 85.0 [62.4 to 95.1] | 70.0 [47.3 to 85.9]

4. Primary Outcome: Median Colony Forming Units Per mL Treatment vs Control
Description: Samples taken from treatment arm and control arm after chlorhexidine (CHX) preparation on both sides.
Time Frame: up to 2 days
Measure: Median (Inter-Quartile Range); unit: CFU/mL
Arm/Group | Blue Light Therapy | 5% Topical Benzoyl Peroxide Gel | Light and Gel
Number analyzed (Participants) | 20 | 20 | 20
CFU/mL
  Treatment plus CHX Arm | 50000 [17000 to 247000] | 2000 [2000 to 2000] | 2000 [2000 to 11300]
  Control Arm after CHX | 108000 [4000 to 254000] | 41500 [2000 to 96000] | 20000 [2000 to 258000]

ADVERSE EVENTS:
Time Frame: Participants were contacted at least 1 week following the final research visit to ask for any delayed side effects of treatments, up to 2 weeks on study
Arm/Group | Blue Light Therapy | 5% Topical Benzoyl Peroxide Gel | Light and Gel | Control Shoulder
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/60
Other Adverse Events (participants affected / at risk) | 6/20 | 6/20 | 6/20 | 2/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blue Light Therapy (N=20) | 5% Topical Benzoyl Peroxide Gel (N=20) | Light and Gel (N=20) | Control Shoulder (N=60)
Itching or Burning (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Skin Dryness, Peeling, or Flaking (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 1
bleaching of clothing (Product Issues) | 0 | 2 | 0 | 0
Erythema (Injury, poisoning and procedural complications) | 3 | 2 | 4 | 1 — transient erythema at application site
Hyperpigmentation (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 — transient hyperpigmentation
Warmth at Treatment Site (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT04300010/Prot_SAP_001.pdf